CLINICAL TRIAL: NCT01790269
Title: Monitoring Natural Killer Cells in Multiple Sclerosis Patients Treated With Fingolimod: a Monocentric, Prospective, One Year, Baseline-to-treatment, Open-label Single Group Pilot Trial
Brief Title: Monitoring Natural Killer Cells in Multiple Sclerosis Patients Treated With Fingolimod
Status: Terminated | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Dr. Carmen Infante-Duarte (Unknown)
Responsible Party: Principal Investigator, Jan-Markus Dörr, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: NKcells Gilenya®-treated MS
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Relapsing-Remitting Multiple Sclerosis; NK cells; Fingolimod
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fingolimod treated patients: Indication for on-label treatment with fingolimod (Gilenya®) according to the current approval

SUMMARY:
Data on fingolimod effects on NK cells are so far conflicting. A longitudinal study on fingolimod treated kidney transplant patients showed that NK cells were not influenced in any of the treatment groups. However, more recent reports indicate an increased frequency of NK cells in peripheral blood and CSF of MS patients treated with fingolimod and a relative reduction of immature CD56bright NK cells in fingolimod-treated MS patients. It has been demonstrated that the expression of NK cell relevant sphingosine 1-phosphate (S1P) receptors seems to increase during NK cell maturation. Thus, different NK cell sub-types may response differently to S1P-receptor agonist such as fingolimod.

Therefore, the investigators aim to investigate longitudinally (baseline vs. treatment) the effects of fingolimod on NK cell maturation/differentiation.

DETAILED DESCRIPTION:
In the past decade, it has become evident that natural killer (NK) cells are more than simply killers and seem to be involved in the regulation of autoimmune conditions such as Multiple Sclerosis (MS). Yet, the complexity of NK cell activation and maturation is only now being understood. Several recent publications have reported on markers characterizing different stages of human NK cell maturation/ differentiation, including CD27, CD62L, CD94 and CD57. In our more recent study, the investigators demonstrated that the chemokine receptor CX3CR1 represents an additional marker for NK cells, which in conjunction with other novel markers, serves to delineate the sequential stages of human NK cell differentiation. CX3CR1 has been suggested to be essential for the protective effects of NK cells in the animal model of MS. In this context, the investigators previously reported on the correlation of the frequency of circulating CX3CR1-positive NK cells with disease activity in patients with MS. Moreover, our unpublished data indicates an association of genetic variation in NK cell-related genes and response to IFN-beta treatment. Thus, it appears that NK cells (or at least certain NK cell fractions) may be not only protective in MS but also mediators of therapeutic benefits.

Fingolimod (GILENYA®) is a modulator of the sphingosine 1-phosphate receptor (S1P-receptors) indicated for the treatment of patients with relapsing forms of MS to reduce the frequency of clinical relapses. Gilenya® is licensed in Germany since April 2011 as an escalation therapy for patients with highly active RRMS.

Data on fingolimod effects on NK cells are so far conflicting. A longitudinal study on fingolimod treated kidney transplant patients showed that NK cells were not influenced in any of the treatment groups. However, more recent reports indicate an increased frequency of NK cells in peripheral blood and CSF of MS patients treated with fingolimod and a relative reduction of immature CD56bright NK cells in fingolimod-treated MS patients. However, this latter study exclusively compared frequencies of NK cells in untreated MS patients and patients treated with fingolimod, while longitudinal intraindividual data during treatment was not presented.

Moreover, these two studies have not considered the potential diverse effects of fingolimod on different NK cells subpopulations. It has been demonstrated that the expression of NK cell relevant sphingosine 1-phosphate (S1P) receptors seems to increase during NK cell maturation. Thus, different NK cell sub-types may response differently to S1P-receptor agonist such as fingolimod.

Therefore, the investigators aim to investigate longitudinally (baseline vs. treatment) the effects of fingolimod on NK cell maturation/differentiation.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of RRMS according to the 2010 revised McDonald criteria (Polman et al., 2011)
* 18 to 64 years old
* Indication for on-label treatment with fingolimod (Gilenya®) ac-cording to the current approval
* EDSS score ≤ 6,0
* Neurological stable with no evidence of relapse or corticosteroid treatment within 30 days prior to screening
* Ability to provide written informed consent
* Highly effective contraception (Pearl Index < 1), reliable abstinence from any heterosexual relationships, or sterilization of the only partner in women of childbearing potential
* Negative pregnancy test (HCG rapid test in the urine) at screening and baseline in women of childbearing potential

Exclusion Criteria:

* Patients with MS manifestations other than RRMS
* Patients with known contraindications to Gilenya® according to the current "Fachinformation", in particular
* Immunodeficiency syndrome
* Increased risk of opportunistic infections
* Severe active or chronic active infections (hepatitis, tuberculosis)
* History or presence of malignancy (other than localized basal or squamous cell carcinoma of the skin). Severe liver dysfunction (Child Pugh C)
* Hypersensitivity against active or any other compound of study medication
* 2nd degree Mobitz Type II or higher degree AV block, Sick-sinus syndrome, or Sinuatrial heart block, Significant QT prolongation (QTc>470 msec (female) or >450 msec (males))
* History of symptomatic bradycardia or recurrent syncope, known ischaemic heart disease, cerebrovascular disease, history of myocardial infarction, hypokalaemia, congestive heart failure, history of cardiac arrest, uncontrolled hypertension, or severe sleep apnea. Patients with clinically significant liver, kidney or bone marrow dysfunction, defined by the following laboratory values at the time of screening:
* HB <8.5 g / dl
* WBC <2.5 / nl
* platelets <100/nl
* creatinine clearance by Cockroft-Gault formula: Cl <110ml/min (men) and Cl <95ml/min (women), from age of 30 limit drops 10ml/min per decade
* AST / ALT> 3.5 times higher than the upper reference value
* bilirubin > 2.0 mg / dl
* Patients without a history of varicella or without vaccination against varicella zoster virus (VZV) and VZV negative antibody serology
* Pregnancy or lactation
* Participation in another interventional clinical trial within the last 3 months prior to baseline or during the study period
* Treatment with Natalizumab within the last 3 months prior to baseline, treatment with mitoxantrone, azathioprine or any other immunosuppressive drugs except prednisolone within the last 6 months prior to baseline.
* Patients receiving antiarrythmics class Ia (e.g. quinidine, disopyramide) or class III (e.g. amiodarone, sotalol) or beta blockers. Patients receiving heart rate lowering calcium channel blockers (e.g. verapamil, diltiazem or ivabradine) or other sub-stances which may decrease heart rate (e.g. digoxin, anticholinesteratic agents or pilocarpine).
* Medical, psychiatric or other conditions that limit the patient' s ability to understand the patient's information, to give informed consent or to follow the study protocol
* Lack of consent to the storage and analysis of pseudonymous data in the context of the clinical trial
* Prisoners or patients that are housed in an judicial institution

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Definite diagnosis of Relapsing-Remitting Multiple Sclerosis according to the 2010 revised McDonald criteria (Polman et al., 2011)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Status of NK cell maturation | Baseline to (12 months) treatment
  Status of NK cell maturation, defined as the ratio immature NK cells / total NK cells (percentage), before fingolimod treatment vs. after 12 months of treatment (V4). The maturation status is determined by the expression of certain cell surface markers which can be evaluated by flow cytometry.

SECONDARY OUTCOMES:
NK cell frequency | Baseline, +1 mo, +3 mo, +6 mo, +12 mo
  NK cell frequency at all time points (determined by flow cytometry)
Percentage immature NK cells/total NK cells | Baseline, +1 mo, +3 mo, +6 mo, +12 mo
  Percentage immature NK cells/total NK cells at all time points
NK cell activation | Baseline, +1 mo, +3 mo, +6 mo, +12 mo
  NK cell activation (expression of certain cell surface markers determined by flow cytometry) at all time points
NK cell maturation and activation | Baseline, +1 mo, +3 mo, +6 mo, +12 mo
  NK cell maturation and activation in relation to clinically detectable therapeutic effect (determined a) by annual relapse rate over study period vs. annualized relapse rate in the preceding two years; and b) by the development of disability (determined by Expanded Disability Status Scale (EDSS) during treatment with fingolimod)
NK cell cytotoxicity and the cytokine production | Baseline, +1 mo, +3 mo, +6 mo, +12 mo
  NK cell cytotoxicity and the cytokine production (IL-15, IL-13, IL-5, GM-CSF, IFN-gamma)

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Markus Dörr, MD, Principal Investigator — Charite Universitätsmedizin Berlin
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- See also: Related Info — http://www.ncrc.de